CLINICAL TRIAL: NCT00704860
Title: Treatment-Resistant Depression, Hippocampus Atrophy and Serotonin Genetic Polymorphism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Pierre Blier, MD, Ph.D., University of Ottawa Institute of Mental Health Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB- 200506
Record Dates: First submitted 2008-06-18; First posted 2008-06-25 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2009-02

CONDITIONS: Major Depression
Keywords: healthy volunteers treatment resistant major depression hippocampus atrophy MRI serotonin genotyping
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TR (Experimental): TR- Subjects defined as having treatment resistant depression, who have failed at least 2 adequate trials of an antidepressant. Subjects will be treated in an open label trial for their depression, with the goal of sustained remission.
  Interventions: Other: Open label pharmacotherapy

INTERVENTIONS:
Other: Open label pharmacotherapy — Dosage and drug types change based on patients need and response.
  doxepin, clomipramine, amoxapine, amitriptyline, maprotiline, desipramine, nortriptyline, trimipramine, imipramine, protriptyline, isocarboxazid, phenelzine, tranylcypromine, moclobemide, fluvoxamine, paroxetine, fluoxetine, sertraline, citalopram, escitalopram, venlafaxine, atomoxetine, pramipexole, bromocriptine, quetiapine, clozapine, olanzapine, ziprasidone, aripiprazole, paliperidone, Risperidone, bupropion, mirtazapine, pindolol, topiramate, trazodone, Lithium,
  Other Names: All classes of antidepressants, based on patient need

SUMMARY:
Reduction of volume of the hippocampus has been associated with major depression in many studies. It has been suggested that antidepressants may protect against hippocampus volume loss in humans associated with multiple episodes of depression and may also reverse the reduction of volume caused by the depression. In addition, genetic markers for serotonin are implicated with depression, and may be an indication of reduced response to antidepressant treatments.

This study aims to enroll patients who are defined as having treatment resistant depression (no remission after at least 2 treatments trials with an antidepressant). They will receive an MRI scan at the initial visit and either 6 months after sustained remission or 12 months after they enter the study for non-remitters. They will also be asked to give a blood sample for genotyping. They will be matched by age and handedness to healthy volunteers with no personal history of depression who will also receive an MRI scan and genotyping.

The first aim is to compare hippocampal volume of depressed subjects to healthy controls. It is anticipated that subjects will initially have smaller hippocampal volume but of those who sustain remission, there will be a small increase in hippocampal volume. It is also anticipated that specific genetic markers will be related to individuals response to antidepressant treatments.

DETAILED DESCRIPTION:
Individuals who are defined as having treatment-resistant major depression (failure of at least 2 trials of an antidepressant at an adequate dose) and currently meet DSM-IV criteria for depression qualify for this study. At the initial visit, each subject is given an MRI in order to perform a volumetric analysis of their hippocampus and a blood sample is taken in order to determine their genotype for the 5-HT1a(serotonin) promoter. Each patient is then aggressively treated (open label) for depression with the goal of remission. A second MRI scan is completed 6 months after sustained remission or 12 months from baseline if remission is not met or sustained.

The investigators will select healthy volunteer controls with no personal or first relative history of depression and match with the subjects based on age and handedness. Genotyping and and MRI scan will be performed on the healthy subjects in order to compare all parameters.

Hypothesis: It is anticipated that the hippocampal volume will be smaller than those of matched controls. It is also anticipated that the Homozygous G(-1019) genotype will be more prevalent in the patient group than in the healthy subjects.

In addition, it is hypothesized that the investigators should find a small increase in hippocampal volume after long-term treatment. Also, most non-responders will be of homozygous G(-1019) 5-HT1a genotype and will have the greatest degree of hippocampal atrophy. Moreover, it is hypothesized that patients carrying a long allele of 5-HTTLPR polymorphism for 5-HTT might show a better response to antidepressants in general. Finally, it is anticipated that the TPH*A variant of the gene coding for tryptophan hydroxylase will be associated with poorer outcome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between ages of 18 to 65 years of age.
* A diagnosis of Major Depression according to the DSM-IV criteria
* Failing to achieve remission while receiving at least two different antidepressants at adequate dosage for at least 6 weeks.
* Initial score of at least 18 on the HAMD-17 item rating scale

Exclusion Criteria:

* A diagnosis of substance abuse or dependence in the last 6 months or a lifetime diagnosis of substance abuse according to the DSM-IV criteria, elicited by inquiry.
* A diagnosis of post-traumatic stress disorder, schizophrenia, schizo-affective disorder and other psychotic disorders, anorexia nervosa or a history of a manic or mixed episode
* Major medical illnesses including endocrine and neurological disorders, as well as a history of significant head trauma
* Exposure to oral or intravenous steroids
* Contraindications to magnetic resonance imaging
* An IQ less than 80

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-02; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Sustained Remission from Depression and Hippocampal Atrophy | 6 months

SECONDARY OUTCOMES:
5-HT1a Genetic Markers | Baseline Visit

CONTACTS AND LOCATIONS:
Overall Officials: Pierre M Blier, MD, Ph.D, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa Institute of Mental Health Research, Ottawa, Ontario, Canada

REFERENCES:
- See also: University of Ottawa Institute of Mental Health research homepage — http://www.imhr.ca